CLINICAL TRIAL: NCT02566902
Title: Comparison of Breath-Enhanced and T-Piece Nebulizers in Children With Acute Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seton Healthcare Family (Other)
Collaborators: University of Texas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR-15-047
Record Dates: First submitted 2015-09-24; First posted 2015-10-02 (Estimated); Results first posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- T-piece Nebulizer (Active Comparator): Pre-treatment spirometry measurement will be performed, intervention with a one time 5mg nebulized albuterol treatment will be administered with the experimental "T-piece Nebulizer" (Hudson RCI® Micro Mist® nebulizer Teleflex Medical®, Research Triangle Park, NJ). Treatment will be administered over 10 minutes. Following this therapy, post-treatment spirometry measurement will be performed.
  Interventions: Device: T-Piece Nebulizer; Drug: Albuterol; Procedure: Pre-Treatment Spirometry Measurement; Procedure: Post-Treatment Spirometry Measurement
- Breath-Enhanced Nebulizer (Experimental): Pre-treatment spirometry measurement will be performed, intervention with a one time 5mg nebulized albuterol treatment will be administered with the experimental "Breath-Enhanced Nebulizer" (NebuTech® HDN®, Breath-Enhanced High Density Jet Nebulizer Salter Labs®, Arvin, CA). Treatment will be administered over 10 minutes. Following this therapy, post-treatment spirometry measurement will be performed.
  Interventions: Device: Breath-Enhanced Nebulizer; Drug: Albuterol; Procedure: Pre-Treatment Spirometry Measurement; Procedure: Post-Treatment Spirometry Measurement

INTERVENTIONS:
Device: T-Piece Nebulizer — Albuterol treatment administered with Hudson RCI® Micro Mist® nebulizer (Teleflex Medical®, Research Triangle Park, NJ)
  Arms: T-piece Nebulizer
Device: Breath-Enhanced Nebulizer — Albuterol treatment administered with NebuTech® HDN®, Breath-Enhanced High Density Jet Nebulizer (Salter Labs®, Arvin, CA)
  Arms: Breath-Enhanced Nebulizer
Drug: Albuterol — One time 5mg nebulized albuterol treatment given with one of two devices over 10 minutes.
  Other Names: albuterol sulfate
Procedure: Pre-Treatment Spirometry Measurement — Bedside spirometry measurements taken prior to albuterol therapy using ndd® EasyOne Plus® spirometer.
Procedure: Post-Treatment Spirometry Measurement — Bedside spirometry measurements taken after albuterol therapy using ndd® EasyOne Plus® spirometer.

SUMMARY:
This is a blinded observer randomized controlled trial comparing two nebulizer devices. The objective of this study is to evaluate the efficacy of two different nebulizers.

DETAILED DESCRIPTION:
The investigators hypothesize that albuterol delivered with a breath-enhanced nebulizer will lead to statistically greater improvement in FEV1 when compared to an equivalent dose delivered via a standard t-piece nebulizer. The primary aim will be to study changes in forced expiratory volume in one second (FEV1) in patients presenting to an urban pediatric emergency department with a moderate to severe acute asthma exacerbation when utilizing these two nebulizers. Secondary aims will include evaluation of hospital admission rates, emergency department (ED) length of stay (LOS), changes in asthma severity scores, vital sign changes, medication side effects, and total quantity of albuterol given in the ED. A distal aim of the study will be to perform a cost analysis; though the investigators will likely need further clinical trials utilizing multiple dose administration in order to accurately analyze cost.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 6 years and < 18 years
* History of physician diagnosed asthma
* Presenting to ED with breathing difficulty or cough
* Initial FEV1 25%-70% predicted
* Parent or guardian speaks English or Spanish.

Exclusion Criteria:

* Pediatric Asthma Score of 0
* Pregnancy or breast-feeding
* Immediate resuscitation required
* Chronic lung disease (other than asthma)
* Congenital heart disease
* Neuromuscular disease
* Suspected intrathoracic foreign body
* Allergy or other contraindication to study medication

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 118 (Actual)
Dates: Start 2015-10; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Wilkinson, MD, Principal Investigator — Seton Healthcare Family
Locations (1):
- Dell Children's Medical Center, Emergency Department, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cates CJ, Welsh EJ, Rowe BH. Holding chambers (spacers) versus nebulisers for beta-agonist treatment of acute asthma. Cochrane Database Syst Rev. 2013 Sep 13;2013(9):CD000052. doi: 10.1002/14651858.CD000052.pub3. PMID 24037768
- [Background] Tien I, Dorfman D, Kastner B, Bauchner H. Metered-dose inhaler: the emergency department orphan. Arch Pediatr Adolesc Med. 2001 Dec;155(12):1335-9. doi: 10.1001/archpedi.155.12.1335. PMID 11732952
- [Background] Mason N, Roberts N, Yard N, Partridge MR. Nebulisers or spacers for the administration of bronchodilators to those with asthma attending emergency departments? Respir Med. 2008 Jul;102(7):993-8. doi: 10.1016/j.rmed.2008.02.009. Epub 2008 Apr 18. PMID 18396026
- [Background] Osmond MH, Gazarian M, Henry RL, Clifford TJ, Tetzlaff J; PERC Spacer Study Group. Barriers to metered-dose inhaler/spacer use in Canadian pediatric emergency departments: a national survey. Acad Emerg Med. 2007 Nov;14(11):1106-13. doi: 10.1197/j.aem.2007.05.009. Epub 2007 Aug 15. PMID 17699806
- [Background] Scott SD, Osmond MH, O'Leary KA, Graham ID, Grimshaw J, Klassen T; Pediatric Emergency Research Canada (PERC) MDI/spacer Study Group. Barriers and supports to implementation of MDI/spacer use in nine Canadian pediatric emergency departments: a qualitative study. Implement Sci. 2009 Oct 13;4:65. doi: 10.1186/1748-5908-4-65. PMID 19828086
- [Background] Mandelberg A, Tsehori S, Houri S, Gilad E, Morag B, Priel IE. Is nebulized aerosol treatment necessary in the pediatric emergency department? Chest. 2000 May;117(5):1309-13. doi: 10.1378/chest.117.5.1309. PMID 10807815
- [Background] Newnham DM, Lipworth BJ. Nebuliser performance, pharmacokinetics, airways and systemic effects of salbutamol given via a novel nebuliser delivery system ("Ventstream"). Thorax. 1994 Aug;49(8):762-70. doi: 10.1136/thx.49.8.762. PMID 8091320
- [Background] Newman SP, Pitcairn GR, Hooper G, Knoch M. Efficient drug delivery to the lungs from a continuously operated open-vent nebulizer and low pressure compressor system. Eur Respir J. 1994 Jun;7(6):1177-81. PMID 7925889
- [Background] Devadason SG, Everard ML, Linto JM, Le Souef PN. Comparison of drug delivery from conventional versus "Venturi" nebulizers. Eur Respir J. 1997 Nov;10(11):2479-83. doi: 10.1183/09031936.97.10112479. PMID 9426082
- [Background] Ho SL, Kwong WT, O'Drowsky L, Coates AL. Evaluation of four breath-enhanced nebulizers for home use. J Aerosol Med. 2001 Winter;14(4):467-75. doi: 10.1089/08942680152744677. PMID 11791687
- [Background] Rubin BK, Fink JB. The delivery of inhaled medication to the young child. Pediatr Clin North Am. 2003 Jun;50(3):717-31. doi: 10.1016/s0031-3955(03)00049-x. PMID 12877243
- [Background] Hess DR. Aerosol delivery devices in the treatment of asthma. Respir Care. 2008 Jun;53(6):699-723; discussion 723-5. PMID 18501026
- [Background] Sabato K, Ward P, Hawk W, Gildengorin V, Asselin JM. Randomized controlled trial of a breath-actuated nebulizer in pediatric asthma patients in the emergency department. Respir Care. 2011 Jun;56(6):761-70. doi: 10.4187/respcare.00142. Epub 2011 Feb 11. PMID 21333060
- [Background] Lin YZ, Huang FY. Comparison of breath-actuated and conventional constant-flow jet nebulizers in treating acute asthmatic children. Acta Paediatr Taiwan. 2004 Mar-Apr;45(2):73-6. PMID 15335114
- [Background] Colacone A, Afilalo M, Wolkove N, Kreisman H. A comparison of albuterol administered by metered dose inhaler (and holding chamber) or wet nebulizer in acute asthma. Chest. 1993 Sep;104(3):835-41. doi: 10.1378/chest.104.3.835. PMID 8365298
- [Background] Schuh S, Johnson DW, Stephens D, Callahan S, Winders P, Canny GJ. Comparison of albuterol delivered by a metered dose inhaler with spacer versus a nebulizer in children with mild acute asthma. J Pediatr. 1999 Jul;135(1):22-7. doi: 10.1016/s0022-3476(99)70322-7. PMID 10393599
- [Background] Wilkinson M, Bulloch B, Garcia-Filion P, Keahey L. Efficacy of racemic albuterol versus levalbuterol used as a continuous nebulization for the treatment of acute asthma exacerbations: a randomized, double-blind, clinical trial. J Asthma. 2011 Mar;48(2):188-93. doi: 10.3109/02770903.2011.554939. Epub 2011 Jan 29. PMID 21275850
- [Background] Aggarwal AN, Gupta D, Jindal SK. The relationship between FEV1 and peak expiratory flow in patients with airways obstruction is poor. Chest. 2006 Nov;130(5):1454-61. doi: 10.1378/chest.130.5.1454. PMID 17099024
- [Background] Eid N, Yandell B, Howell L, Eddy M, Sheikh S. Can peak expiratory flow predict airflow obstruction in children with asthma? Pediatrics. 2000 Feb;105(2):354-8. doi: 10.1542/peds.105.2.354. PMID 10654955
- [Background] Schneider WV, Bulloch B, Wilkinson M, Garcia-Filion P, Keahey L, Hostetler M. Utility of portable spirometry in a pediatric emergency department in children with acute exacerbation of asthma. J Asthma. 2011 Apr;48(3):248-52. doi: 10.3109/02770903.2011.555036. Epub 2011 Feb 21. PMID 21332428
- [Background] Qureshi F, Pestian J, Davis P, Zaritsky A. Effect of nebulized ipratropium on the hospitalization rates of children with asthma. N Engl J Med. 1998 Oct 8;339(15):1030-5. doi: 10.1056/NEJM199810083391503. PMID 9761804
- [Background] Gorelick MH, Stevens MW, Schultz TR, Scribano PV. Performance of a novel clinical score, the Pediatric Asthma Severity Score (PASS), in the evaluation of acute asthma. Acad Emerg Med. 2004 Jan;11(1):10-8. doi: 10.1197/j.aem.2003.07.015. PMID 14709423
- [Background] Barr RG, Stemple KJ, Mesia-Vela S, Basner RC, Derk SJ, Henneberger PK, Milton DK, Taveras B. Reproducibility and validity of a handheld spirometer. Respir Care. 2008 Apr;53(4):433-41. PMID 18364054
- [Background] Standardization of Spirometry, 1994 Update. American Thoracic Society. Am J Respir Crit Care Med. 1995 Sep;152(3):1107-36. doi: 10.1164/ajrccm.152.3.7663792. No abstract available.
- [Background] Gorelick MH, Stevens MW, Schultz T, Scribano PV. Difficulty in obtaining peak expiratory flow measurements in children with acute asthma. Pediatr Emerg Care. 2004 Jan;20(1):22-6. doi: 10.1097/01.pec.0000106239.72265.16. PMID 14716161
- [Derived] Gardiner MA, Wilkinson MH. Interrater Reliability of the Pediatric Asthma Score. Pediatr Emerg Care. 2022 Apr 1;38(4):143-146. doi: 10.1097/PEC.0000000000002556. PMID 34693935
- [Derived] Gardiner MA, Wilkinson MH. Randomized Clinical Trial Comparing Breath-Enhanced to Conventional Nebulizers in the Treatment of Children with Acute Asthma. J Pediatr. 2019 Jan;204:245-249.e2. doi: 10.1016/j.jpeds.2018.08.083. Epub 2018 Nov 2. PMID 30392872
- See also: American Lung Association, Epidemiology and Statistics Unit. Trends in Asthma Morbidity and Mortality. 2012 — https://www.lung.org/research/trends-in-lung-disease/asthma-trends-brief/trends-and-burden

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | T-piece Nebulizer | Breath-Enhanced Nebulizer
Started | 60 | 58
Completed | 58 | 57
Not Completed | 2 | 1
Not completed — Protocol Violation | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | T-piece Nebulizer | Breath-Enhanced Nebulizer | Total
Number analyzed (Participants) | 58 | 57 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.8 (2.6) | 10.1 (3.0) | 9.98 (2.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 30 | 51
  Male | 37 | 27 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 33 | 63
  Not Hispanic or Latino | 28 | 24 | 52
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 58 | 57 | 115
Baseline Asthma Severity [Count of Participants; unit: Participants]
  Mild Intermittent | 20 | 27 | 47
  Mild Persistent | 11 | 12 | 23
  Moderate Persistent | 20 | 14 | 34
  Severe Persistent | 7 | 4 | 11
Weight (kg) [Mean (Standard Deviation); unit: kilograms] | 39.5 (16.4) | 41.1 (16.5) | 40.7 (16.5)
Duration of symptoms (days) [Median (Inter-Quartile Range); unit: days] | 2 [1 to 3] | 2 [2 to 3] | 2 [1 to 3]
Initial RR (bpm) [Mean (Standard Deviation); unit: breaths/min] | 28.1 (9.4) | 28.9 (7.6) | 28.4 (8.5)
Initial O2 [Mean (Standard Deviation); unit: %saturation] | 96.0 (2.1) | 95.7 (2.6) | 95.8 (2.4)
Initial PAS score [Median (Inter-Quartile Range); unit: units on a scale] — Determined by examination and auscultation of lungs prior to albuterol administration.
  PAS score is on a scale of 0-10 which is a sum of five separate sub-scores each on a scale of 0-2. The five sub-scores are:
  1. Respiratory rate (6-12yr/>12yr): <=26/23 (0), 27-30/24-27 (1), >31/28 (2)
  2. Oxygenation: >95% (0), 90-95 (1), <90 (2)
  3. Auscultation: clear/end expiratory wheeze (0), expiratory wheeze (1), biphasic wheeze/diminished (2)
  4. Work of Breathing (accessory muscles): <= 1 (0), 2 (1), >=3 (2)
  5. Dyspnea: Full sentences (0), Partial sentences (1), Single words (2)
  units on a scale | 4 [3 to 5] | 4 [2 to 5] | 4 [3 to 5]
Initial PASS score [Median (Inter-Quartile Range); unit: units on a scale] — Determined by examination and auscultation of lungs prior to albuterol administration.
  PASS is a total score on a scale of 0-6 which is calculated as a sum of three sub-scores, each on a scale of 0-2. The sub-scores are:
  1. Wheezing: None or Mild (0), Moderate (1), Severe wheezing or absent wheezing due to poor air exchange (2)
  2. Work of breathing (accessory muscle use or retractions): None or mild (0), Moderate (1), Severe (2)
  3. Prolonged expiration: Normal or mildly prolonged (0), moderately prolonged (1), severely prolonged (2)
  units on a scale | 2 [2 to 3] | 2 [1 to 3] | 2 [1 to 3]
Initial FEV1 (% predicted) [Mean (Standard Deviation); unit: %predicted] | 39.4 (13.4) | 42 (14.8) | 40.5 (14.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in FEV1 (% Predicted)
Description: Pre-treatment spirometry measurement assessed at the time of study enrollment. Post-treatment spirometry measurement assessed following the administration of one time 5mg nebulized albuterol sulfate treatment. Assessments taken at baseline (prior to albuterol therapy) and 10 min post-treatment. Change in FEV1 calculated as post-treatment FEV1 minus pre-treatment FEV1
Time Frame: 10 minutes
Population: Eight subjects unable to complete post-treatment spirometry (three in T-piece group, five in breath-enhanced group)
Measure: Mean (95% Confidence Interval); unit: %predicted
Arm/Group | T-piece Nebulizer | Breath-Enhanced Nebulizer
Number analyzed (Participants) | 55 | 52
%predicted | 13.8 [10.5 to 17.2] | 9.1 [6.1 to 12.1]
Statistical Analysis 1: Comparison: T-piece Nebulizer vs Breath-Enhanced Nebulizer; Test type: Superiority; p = 0.04, t-test, 2 sided

2. Secondary Outcome: Change in PAS Score (Points on a Scale)
Description: Based on examination and auscultation of lungs prior to and immediately following albuterol administration.
  PAS score is on a scale of 0-10 which is a sum of five separate sub-scores each on a scale of 0-2. The five sub-scores are:
  1. Respiratory rate (6-12yr/>12yr): <=26/23 (0), 27-30/24-27 (1), >31/28 (2)
  2. Oxygenation: >95% (0), 90-95 (1), <90 (2)
  3. Auscultation: clear/end expiratory wheeze (0), expiratory wheeze (1), biphasic wheeze/diminished (2)
  4. Work of Breathing (accessory muscles): <= 1 (0), 2 (1), >=3 (2)
  5. Dyspnea: Full sentences (0), Partial sentences (1), Single words (2)
  Pre-treatment assessment at the time of study enrollment. Post-treatment assessment following the administration of one time 5mg nebulized albuterol sulfate treatment. Assessments taken at baseline (prior to albuterol therapy) and 10 min post-treatment. Change in PAS calculated as post-treatment PAS minus pre-treatment PAS.
Time Frame: 10 minutes
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | T-piece Nebulizer | Breath-Enhanced Nebulizer
Number analyzed (Participants) | 58 | 57
score on a scale | -1 [-2 to -1] | -2 [-2 to -1]
Statistical Analysis 1: Comparison: T-piece Nebulizer vs Breath-Enhanced Nebulizer; Test type: Superiority; p = 0.29, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in PASS Score (Points on a Scale)
Description: Determined by examination and auscultation of lungs to prior to and immediately following albuterol administration.
  PASS is a total score on a scale of 0-6 which is calculated as a sum of three sub-scores, each on a scale of 0-2. The sub-scores are:
  1. Wheezing: None or Mild (0), Moderate (1), Severe wheezing or absent wheezing due to poor air exchange (2)
  2. Work of breathing (accessory muscle use or retractions): None or mild (0), Moderate (1), Severe (2)
  3. Prolonged expiration: Normal or mildly prolonged (0), moderately prolonged (1), severely prolonged (2)
  Pre-treatment assessment at the time of study enrollment. Post-treatment assessment following the administration of one time 5mg nebulized albuterol sulfate treatment. Assessments taken at baseline (prior to albuterol therapy) and 10 min post-treatment. Change in PASS calculated as post-treatment PASS minus pre-treatment PASS.
Time Frame: 10 minutes
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | T-piece Nebulizer | Breath-Enhanced Nebulizer
Number analyzed (Participants) | 58 | 57
score on a scale | -1 [-1 to 0] | -1 [-1 to 0]
Statistical Analysis 1: Comparison: T-piece Nebulizer vs Breath-Enhanced Nebulizer; Test type: Superiority; p = 0.97, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Percentage of Patients Requiring Inpatient Hospital Admission (% of Subjects)
Description: Admission rate to inpatient hospital will be assessed at the time of Emergency Department disposition which will be approximately 3 hours, but will be assessed up to 24 hours depending on duration of ED stay.
Time Frame: Up to 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | T-piece Nebulizer | Breath-Enhanced Nebulizer
Number analyzed (Participants) | 58 | 57
Participants | 11 | 11
Statistical Analysis 1: Comparison: T-piece Nebulizer vs Breath-Enhanced Nebulizer; Test type: Superiority; p = 0.96, Chi-squared

5. Secondary Outcome: Emergency Department Length of Stay (Minutes)
Description: Total length of stay will be assessed at the time of Emergency Department disposition which will be approximately 3 hours, but will be assessed up to 24 hours depending on duration of ED stay.
Time Frame: Up to 24 hours
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | T-piece Nebulizer | Breath-Enhanced Nebulizer
Number analyzed (Participants) | 58 | 57
minutes | 246.3 [220.4 to 272.3] | 246.2 [220.4 to 272.0]
Statistical Analysis 1: Comparison: T-piece Nebulizer vs Breath-Enhanced Nebulizer; Test type: Superiority; p = 0.99, t-test, 2 sided

6. Secondary Outcome: Percentage of Patients Experiencing Medication Side Effects (%)
Description: Subjects and parents/guardians will be asked whether subjects experienced nausea, vomiting, palpitations, headache, dizziness either during (assessed by non-blinded personnel) or following treatment (assessed by blinded personnel during post-treatment assessment). Subject and parent/guardian will also be asked if any "other" side effects were experienced.
Time Frame: 10 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | T-piece Nebulizer | Breath-Enhanced Nebulizer
Number analyzed (Participants) | 58 | 57
Participants | 5 | 5
Statistical Analysis 1: Comparison: T-piece Nebulizer vs Breath-Enhanced Nebulizer; Test type: Superiority; p = 1.00, Fisher Exact

7. Secondary Outcome: Total Quantity of Albuterol Given in the Emergency Department (mg)
Description: Cumulative dose of albuterol in mg will be assessed at the time of Emergency Department disposition which will be approximately 3 hours, but will be assessed up to 24 hours depending on duration of ED stay.
Time Frame: up to 24 hours
Measure: Mean (95% Confidence Interval); unit: mg
Arm/Group | T-piece Nebulizer | Breath-Enhanced Nebulizer
Number analyzed (Participants) | 58 | 57
mg | 18.2 [14.3 to 22.1] | 18.7 [15.0 to 22.3]

8. Secondary Outcome: Change Respiratory Rate (Breaths Per Minute)
Description: Respiratory rate will be measured by observation and auscultation over 30 seconds prior to and immediately following albuterol administration
  Pre-treatment assessment at the time of study enrollment. Post-treatment assessment following the administration of one time 5mg nebulized albuterol sulfate treatment. Assessments taken at baseline (prior to albuterol therapy) and 10 min post-treatment. Change in respiratory rate calculated as post-treatment respiratory rate minus pre-treatment respiratory rate.
Time Frame: 10 minutes
Measure: Mean (95% Confidence Interval); unit: breaths/min
Arm/Group | T-piece Nebulizer | Breath-Enhanced Nebulizer
Number analyzed (Participants) | 58 | 57
breaths/min | -3.1 [-4.7 to -1.4] | -3.2 [-4.9 to -1.5]

9. Secondary Outcome: Change in Heart Rate (Beats Per Minute)
Description: Blinded research personnel will assess subject's heart rate by auscultation and/or pulse palpation prior to and immediately following albuterol administration.
  Pre-treatment assessment at the time of study enrollment. Post-treatment assessment following the administration of one time 5mg nebulized albuterol sulfate treatment. Assessments taken at baseline (prior to albuterol therapy) and 10 min post-treatment. Change in heart rate calculated as post-treatment heart rate minus pre-treatment heart rate.
Time Frame: 10 minutes
Measure: Mean (95% Confidence Interval); unit: beats per minute
Arm/Group | T-piece Nebulizer | Breath-Enhanced Nebulizer
Number analyzed (Participants) | 58 | 57
beats per minute | 4.34 [0.68 to 8.01] | 15.05 [10.66 to 19.45]

ADVERSE EVENTS:
Time Frame: Duration of emergency department visit until the time of discharge or admission - up to 24 hours.
Arm/Group | T-piece Nebulizer | Breath-Enhanced Nebulizer
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/57
Other Adverse Events (participants affected / at risk) | 5/58 | 5/57
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T-piece Nebulizer (N=58) | Breath-Enhanced Nebulizer (N=57)
Shakiness, Jitteriness (Nervous system disorders) | 2 (2) | 1 (1) — Subjective shakiness or dizziness
Dizziness (Nervous system disorders) | 3 (3) | 2 (2) — Subjective dizziness
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Weakness (Nervous system disorders) | 1 (1) | 0 (0) — Subjective feeling of weakness

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-30): https://cdn.clinicaltrials.gov/large-docs/02/NCT02566902/Prot_SAP_000.pdf